CLINICAL TRIAL: NCT01695863
Title: Phase 4 of Efficacy and Patient Satisfaction of Miralax and Gatorade Versus Movi Prep
Brief Title: Efficacy and Patient Satisfaction of Miralax and Gatorade Versus Movi Prep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 11042705
Record Dates: First submitted 2012-08-10; First posted 2012-09-28 (Estimated); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
Keywords: Miralax with gatorade and dulcolax; Movi pre; Patient satisfaction and efficacy
MeSH Terms: conditions — Colorectal Neoplasms; Patient Satisfaction | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- miralax (Experimental): miralax with dulcolax and gatorade efficacy evaluated by colonoscopy and patient satisfaction evaluated by patient questionnaire
  Interventions: Drug: comparing 2 drugs on their effect on the bowel preparation for colonoscopy
- moviprep split dose (Experimental): Efficacy of split dose moviprep on cleansing colon for colonoscopy and patient satisfaction with the regimen
  Interventions: Drug: comparing 2 drugs on their effect on the bowel preparation for colonoscopy

INTERVENTIONS:
Drug: comparing 2 drugs on their effect on the bowel preparation for colonoscopy — the effects of the drug on the colon preparation for colonoscopy

SUMMARY:
This study will be comparing patient satisfaction, efficacy comparing miralax with gatorade versus Movi Prep for outpatient colonoscopy.

DETAILED DESCRIPTION:
Study is the purpose of evaluating patient satisfaction and at the same time efficacy of the bowel regimen in cleansing the colon

ELIGIBILITY:
Inclusion Criteria:

* outpatient colonoscopy for screening for other Gi related problems

Exclusion Criteria:

* Severe Congestive Heart Failure (CHF),
* Chronic Kidney Disease (CKD),
* less than age 18 or more than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maqsood A Khan, MD, Principal Investigator — Rush University Medical Center; Ali Keshavarzian, MD, Study Chair — RUMC; Michael D Brown, MD, Study Director — RUMC; John losurdo, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Unversity Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Hookey LC, Vanner S. A review of current issues underlying colon cleansing before colonoscopy. Can J Gastroenterol. 2007 Feb;21(2):105-11. doi: 10.1155/2007/634125. PMID 17299615
- [Background] DiPalma JA, Wolff BG, Meagher A, Cleveland Mv. Comparison of reduced volume versus four liters sulfate-free electrolyte lavage solutions for colonoscopy colon cleansing. Am J Gastroenterol. 2003 Oct;98(10):2187-91. doi: 10.1111/j.1572-0241.2003.07690.x. PMID 14572566
- See also: rush university medical center website — http://rush.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 150 patients were recruited and randomized to 75 patients in each arm. Of these, 128 patients arrived for the colonoscopy; therefore eligible to enter the final analysis.
Pre-assignment Details: To be able to enter a recruited patient into analysis, the consented patient must complete their colonoscopy. Of the 150 consented patients, 128 completed their colonoscopy while the remaining 22 did not. Those who did not complete their colonoscopy were excluded from analysis.
Groups:
- Miralax: Miralax with Dulcolax and Gatorade given orally prior to surgery
- Moviprep Split Dose: Split dose Moviprep given orally prior to surgery
Period: Overall Study
Arm/Group | Miralax | Moviprep Split Dose
Started | 62 | 66
Completed | 62 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Miralax: Miralax with Dulcolax and Gatorade given prior to surgery.
- Moviprep Split Dose: Split dose Moviprep on cleansing colon given prior to surgery
- Total: Total of all reporting groups
Arm/Group | Miralax | Moviprep Split Dose | Total
Number analyzed (Participants) | 62 | 66 | 128
Age, Customized [Count of Participants; unit: Participants]
  Age > 18 Years | 62 | 66 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Bowel Prep Efficacy - Boston Bowel Preparation Scale (BBPS)
Description: To assess the bowel prep efficacy in cleansing the colon for colonoscopy - Scale used is the Boston Bowel Preparation Scale (BBPS), Integer Scale from 0-3, where 3 indicated the best outcome and 0 the worst. The BBPS was estimated during the procedure (Colonoscopy) by an endoscopist and a nurse and retrospectively by a second endoscopist postoperatively. Scores were averaged by for each subject by location (Right colon, Transverse colon, and Left colon) and then for each group/arm by location.
Time Frame: Outcome BBPS was measured during surgery for endoscopist #1 and nurse raters and post-operatively (at any time before the end of the study) by endoscopist #2
Population: A few of the outcomes had Missing data since the evaluations were not complete for specific locations by the clinical personnel.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Miralax: Miralax with Dulcolax and Gatorade efficacy evaluated by colonoscopy
- Moviprep Split Dose: Efficacy of split dose moviprep on cleansing colon for colonoscopy
Arm/Group | Miralax | Moviprep Split Dose
Number analyzed (Participants) | 62 | 66
score on a scale
  Right Colon: number analyzed (Participants) | 62 | 65
  Right Colon | 1.79 (0.72) | 2.33 (.89)
  Transverse Colon: number analyzed (Participants) | 61 | 66
  Transverse Colon | 2.06 (0.79) | 2.45 (0.72)
  Left Colon | 2.24 (0.76) | 2.46 (0.70)
Statistical Analysis 1: Comparison: Miralax vs Moviprep Split Dose; Right Colon; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = .54, 95% CI 2-sided [0.269 to 0.816]
Statistical Analysis 2: Comparison: Miralax vs Moviprep Split Dose; Transverse Colon; Test type: Superiority; p = 0.005, t-test, 2 sided; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.122 to 0.655]
Statistical Analysis 3: Comparison: Miralax vs Moviprep Split Dose; Left Colon; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.029 to 0.484]

2. Secondary Outcome: Renal Function Pre and Post Bowel Prep (mg/dL)
Description: Changes in electrolytes pre and post bowel preparation administration. Pre bowel prep measures were taken at study randomization (up to one week before surgery) and post bowel prep measures were taken prior to the procedure (less than 5 hours before start of procedure on day of procedure). Change is electrolytes are presented as pre bowel prep value minus post bowel prep value but prior to procedure (Pre-Post). Units = Milligrams/deciLiter (mg/dL)
Time Frame: Pre bowel prep measures were taken at study randomization (up to one week before surgery) and post bowel prep measures were taken prior to the procedure (less than 5 hours before start of procedure on day of procedure).
Measure: Mean (Standard Deviation); unit: Milligram per deciLiter (mg/dL)
Groups:
- Miralax: Miralax with Dulcolax and Gatorade - Given Orally
- Moviprep Split Dose: Split dose Moviprep - Given Orally
Arm/Group | Miralax | Moviprep Split Dose
Number analyzed (Participants) | 62 | 66
Milligram per deciLiter (mg/dL)
  Calcium | 0.18 (.53) | 0.02 (.53)
  Glucose | 1.41 (45.44) | 3.44 (45.44)
  Blood Urea Nitrogen | 3.44 (4.72) | 3.00 (4.72)
  Creatinine | -0.01 (0.14) | -0.02 (0.14)
Statistical Analysis 1: Comparison: Miralax vs Moviprep Split Dose; Calcium; Test type: Superiority; p = 0.093, t-test, 2 sided; Mean Difference (Final Values) = -0.16
Statistical Analysis 2: Comparison: Miralax vs Moviprep Split Dose; Glucose; Test type: Superiority; p = 0.801, t-test, 2 sided; Mean Difference (Final Values) = 2.03
Statistical Analysis 3: Comparison: Miralax vs Moviprep Split Dose; Blood Urea Nitrogen; Test type: Superiority; p = 0.599, t-test, 2 sided; Mean Difference (Final Values) = -0.44
Statistical Analysis 4: Comparison: Miralax vs Moviprep Split Dose; Creatinine; Test type: Superiority; p = 0.696, t-test, 2 sided; Mean Difference (Final Values) = -0.01
Statistical Analysis 5: Comparison: Miralax vs Moviprep Split Dose; Sodium; Test type: Superiority; p = .042, t-test, 2 sided; Mean Difference (Final Values) = -1.19
Statistical Analysis 6: Comparison: Miralax vs Moviprep Split Dose; Potassium; Test type: Superiority; p = 0.596, t-test, 2 sided; Mean Difference (Final Values) = 0.07
Statistical Analysis 7: Comparison: Miralax vs Moviprep Split Dose; Chloride; Test type: Superiority; p = 0.107, t-test, 2 sided; Mean Difference (Final Values) = -0.98
Statistical Analysis 8: Comparison: Miralax vs Moviprep Split Dose; Bicarbonate; Test type: Superiority; p = 0.351, t-test, 2 sided; Mean Difference (Final Values) = 0.71

3. Other Pre Specified Outcome: Non-Serious Adverse Events on Self Report Scale
Description: Non-Serious Adverse Events on self report scale - 5 point scale from "No Complaints (0)" to "Very Severe (4)" with 4 indicating the worst outcome and 0 the best.
Time Frame: During Bowel Preparation (Pre-Operative)
Population: These are self-report measures and not all subject submitted or complete the self report measures. Of 62 in the Miralax condition 43 retuned the self-report questionnaire (19 did not) and of 66 in the Moviprep condition 51 returned the self-report questionnaire (15 did not).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Miralax: miralax with dulcolax and gatorade
- Moviprep Split Dose: Split dose Moviprep given orally
Arm/Group | Miralax | Moviprep Split Dose
Number analyzed (Participants) | 43 | 51
score on a scale
  Nausea | 0.3590 (0.77) | 0.3152 (0.61)
  Vomiting | 0.2821 (0.85) | 0.0000 (0.0000)
  Bloating | 0.6667 (0.89) | 0.4565 (0.72)
  Abdominal pain or cramping | 0.359 (0.66) | 0.3043 (0.66)
  Ability to complete entire prep | 1.878 (0.39) | 1.8511 (0.46)
  Difficulty/Inconvenience in completing prep | 0.6098 (0.80) | 0.6596 (0.75)
Statistical Analysis 1: Comparison: Miralax vs Moviprep Split Dose; Nausea; Test type: Superiority; p = 0.772, t-test, 2 sided; Mean Difference (Final Values) = -0.0438
Statistical Analysis 2: Comparison: Miralax vs Moviprep Split Dose; Vomiting; Test type: Superiority; p = 0.028, t-test, 2 sided; Mean Difference (Final Values) = -0.2821
Statistical Analysis 3: Comparison: Miralax vs Moviprep Split Dose; Bloating; Test type: Superiority; p = 0.235, t-test, 2 sided; Mean Difference (Final Values) = -0.2102
Statistical Analysis 4: Comparison: Miralax vs Moviprep Split Dose; Abdominal pain or cramping; Test type: Superiority; p = 0.707, t-test, 2 sided; Mean Difference (Final Values) = -0.0547
Statistical Analysis 5: Comparison: Miralax vs Moviprep Split Dose; Ability to complete entire prep; Test type: Superiority; p = 0.773, t-test, 2 sided; Mean Difference (Final Values) = -0.0269
Statistical Analysis 6: Comparison: Miralax vs Moviprep Split Dose; Difficulty/Inconvenience in completing prep; Test type: Superiority; p = 0.766, t-test, 2 sided; Mean Difference (Final Values) = 0.0498

4. Secondary Outcome: Renal Function Pre and Post Bowel Prep - Continued (mmol/L)
Description: Changes in electrolytes pre and post bowel preparation administration. Pre bowel prep measures were taken at study randomization (up to one week before surgery) and post bowel prep measures were taken prior to the procedure (less than 5 hours before start of procedure on day of procedure). Change is electrolytes are presented as pre bowel prep value minus post bowel prep value, but prior to procedure (Pre-Post). Units=Millimoles per Liter (mmol/L)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Miralax | Moviprep Split Dose
Number analyzed (Participants) | 62 | 66
Millimoles per Liter (mmol/L)
  Sodium | 0.27 (3.28) | -0.92 (3.28)
  Potassium | -0.18 (0.74) | -0.11 (0.74)
  Chloride | 0.54 (3.41) | -0.44 (3.41)
  Bicarbonate | 1.43 (4.29) | 2.14 (4.29)

ADVERSE EVENTS:
Time Frame: 8 Months for Adverse Events. For side effects, "Other (Not Including Serious) Adverse Events", the questionnaire for bowl prep solution was given preoperatively and collected before surgery (3 days before surgery to day of surgery).
Description: Adverse events are reported here. Side effects were reported on a self-report scale in the outcomes section and as such the sample sizes were smaller for both groups since some subjects did not complete the questionnaire.
  Of 62 in the Miralax condition 43 retuned the self-report questionnaire (19 did not) and of 66 in the Moviprep condition 51 returned the self-report questionnaire (15 did not).
Groups:
- Miralax: miralax with dulcolax and gatorade Condition
- Moviprep Split Dose: Split dose moviprep Condition
Arm/Group | Miralax | Moviprep Split Dose
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/66
Other Adverse Events (participants affected / at risk) | 22/43 | 28/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Miralax (N=43) | Moviprep Split Dose (N=51)
Nausea (Gastrointestinal disorders) | 12 | 14 — Likert score >0 on 0-4 scale, 0 (No Complaints) to 4 (Very Severe)
Vomiting (Gastrointestinal disorders) | 6 | 0 — Likert score >0 on 0-4 scale, 0 (No Complaints) to 4 (Very Severe)
Bloating (Gastrointestinal disorders) | 22 | 18 — Likert score >0 on 0-4 scale, 0 (No Complaints) to 4 (Very Severe)
Abdominal Pain or Cramping (Gastrointestinal disorders) | 13 | 12 — Likert score >0 on 0-4 scale, 0 (No Complaints) to 4 (Very Severe)
Inability to Complete Prep (Product Issues) | 1 | 2 — Likert score >0 on 0-4 scale, 0 (No Complaints) to 4 (Very Severe)
Difficulty in Completing Prep (Product Issues) | 21 | 28 — Likert score >0 on 0-4 scale, 0 (No Complaints) to 4 (Very Severe)

LIMITATIONS AND CAVEATS:
No systematic recording of incidence for non-serious adverse events were collected by study personnel or subjects, so details on event occurrence cannot be provided. Adverse events on a self-report scale of severity are recorded the table names: "Non-Serious Adverse Events on Self Report Scale" and provide an index of the perceived impact of non-serious adverse events on the subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes